CLINICAL TRIAL: NCT02393534
Title: The Feasibility of Replacing Follow-up Visits With Telephone Calls in Primary Care: A Randomized Clinical Trial
Brief Title: Feasibility of Telephone Follow-up Visits in Primary Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: New York City Health and Hospitals Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 14-01863
Record Dates: First submitted 2015-03-09; First posted 2015-03-19 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: No Specific Condition
Keywords: Primary Care; Health Services Research; Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Eligible patients that are randomized to the usual care arm will have a standard in-person clinic visit with their primary care provider.
- Telephone visit (Experimental): Eligible patients that are randomized to the telephone follow-up arm will have their next medical visit with their primary care provider via a telephone call.
  Interventions: Other: Telephone Visit

INTERVENTIONS:
Other: Telephone Visit — Eligible patients that are randomized to the telephone follow-up arm will have their next medical visit with their primary care provider via a telephone call.
  Arms: Telephone visit

SUMMARY:
Doctors frequently speak with their patients over the telephone. Having a visit with a doctor over the telephone rather than face-to-face can be convenient for patients and allow them to save time and money on transportation and missed time from work. However, some patients may prefer seeing the doctor in person. In this study, we will study two groups of patients - some who have their visits with their doctor over the telephone and some who have them face-to-face. Using surveys and interviews, we will study if the groups differ in their satisfaction with their visit with their doctor after participating in the study for 6 months. We will also look at doctor satisfaction with telephone visits, use of clinic resources and if patients received recommended care such as laboratory tests and vaccines during the study period.

DETAILED DESCRIPTION:
This two arm randomized controlled trial will evaluate the effect of telephone follow-up versus standard in-person follow-up (usual care) on patient satisfaction among a sample of 360 primary care patients followed at the Gouverneur Ambulatory Care Practice. All primary care patients will be considered eligible at the outset. Providers will determine patient's study eligibility at the baseline visit based on the ability to safely follow-up the patient's health issue over the telephone in subsequent visits. Eligible patients that are randomized to the telephone follow-up arm will have their next medical visit with their primary care provider via a telephone call. Eligible patients that are randomized to the usual care arm will have a standard in-person clinic visit with their primary care provider. In both study arms, the timing and frequency of follow-up appointments will be determined by the patient's primary care provider. Regardless of group assignment, outcomes will be assessed at the baseline and 6-month study visit.

ELIGIBILITY:
Inclusion Criteria:

* Have a follow-up issue that can be addressed over the phone (as determined by their provider);
* 18 years of age or older;
* Have a working telephone number; and
* Are English, Spanish, Cantonese or Mandarin-speaking.

Exclusion Criteria:

* Patient refusal or are unable to provide informed consent;
* Currently participate in another clinical trial;
* Have significant psychiatric comorbidity or cognitive impairment that would compromise their ability to participate (as determined by their provider); or
* Plan to discontinue care at the Gouverneur Ambulatory Care Practice within the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Feasibility assessment | 6 months
  Proportion of patients recruited out of the total population and proportion of patients retained at 6 months.

SECONDARY OUTCOMES:
Provider workload | 6 months
  The number of minutes spent in conversation during the telephone visit
Provider workload | 6 months
  The total number of scheduled and unscheduled clinic sessions
Patient Satisfaction | 6 months
  Patient satisfaction assessed with the CG-CAHPS questionnaire. For the purposes of this study we will only use measures related to provider ratings and communication . Semi-structured in-depth interviews will also be conducted with a subsample of patients in the telephone visit arm to elicit their beliefs on the usefulness and appropriateness of telephone visits for their health care needs as well as suggestions for instituting a telephone visit program, and willingness to participate in future telephone visits.

OTHER OUTCOMES:
Provider Satisfaction | 6 months
  Provider satisfaction will be assessed with a Likert-type scale that assesses satisfaction with the telephone medicine program after 6 months of participation. A focus group will also be conducted to elicit providers' opinions beliefs regarding the logistical, organizational, and administrative barriers to conducting telephone follow-up visits, usefulness/suitability of telephone visit to address patient concerns, disadvantages and advantages of using telephone visits, opinions on which patients benefit the most from the service, suggestions for improving the process.
Patient receipt of medical recommendations | 6 months
  Electronic medical records (EMR) will be reviewed to collect data on patient's comorbid conditions, receipt of chronic disease management measures (i.e., blood pressure checks, HbA1c levels), and clinic appointment attendance (i.e., number of visits scheduled with the provider but not attended during the 6-month study period divided by the total number of visits scheduled). Documentation of the receipt of chronic disease management measures (e.g. whether or not patient had recommended blood tests performed) will be used as a proxy for patient adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Schoenthaler, Principal Investigator — NYU School of Medicine
Locations (1):
- Gouverneur TDC, New York, New York, United States